CLINICAL TRIAL: NCT05754840
Title: A Randomized, Double-Blind Tolerability Trial of Cannabinoids for Symptom Management in Children With Cancer: the CAN-PONC Trial
Brief Title: CANnabinoids in Pediatric ONCology
Acronym: CAN-PONC
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Lauren Kelly, Lauren E Kelly PhD, MSc, BMedSci, CCRP, Assistant Professor, Dept. of Pediatrics & Child Health, University of Manitoba Scientific Director, Canadian Childhood Cannabinoid Clinical Trials (www.C4Trials.org), University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CAN-PONC
Record Dates: First submitted 2023-02-13; First posted 2023-03-06 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Childhood Cancer; Cancer
Keywords: cannabinoids; CBD; THC; pediatrics; cannabis
MeSH Terms: conditions — Neoplasms; Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1. High-CBD arm (MPL-001) (Experimental): High-CBD arm (MPL-001) a cannabidiol-enriched cannabis herbal extract which contains a 1:25 ratio of THC:CBD.
  Interventions: Drug: MPL-001
- Arm 2. Medium-CBD arm (MPL-005) (Experimental): Medium-CBD arm (MPL-005) a cannabidiol-enriched cannabis herbal extract which contains a 1:5 ratio of THC:CBD.
  Interventions: Drug: MPL-005
- Arm 3. Balanced arm (MPL-009) (Experimental): Balanced arm (MPL-009) a balanced 1:1 ratio of THC:CBD.
  Interventions: Drug: MPL-009

INTERVENTIONS:
Drug: MPL-001 — High-CBD arm (MPL-001) a cannabidiol-enriched cannabis herbal extract which contains a 1:25 ratio of THC:CBD. The MPL-001 oil is produced by MediPharm Labs, each ml contains 50mg CBD and 2mg THC.
  Arms: Arm 1. High-CBD arm (MPL-001)
Drug: MPL-005 — Medium-CBD arm (MPL-005) a cannabidiol-enriched cannabis herbal extract which contains a 1:5 ratio of THC:CBD. The MPL-005 oil is produced by MediPharm Labs, each ml contains 25mg CBD and 5mg THC.
  Arms: Arm 2. Medium-CBD arm (MPL-005)
Drug: MPL-009 — Balanced arm (MPL-009) a balanced 1:1 ratio of THC:CBD. The MPL-009 oil is produced by MediPharm Labs, each ml contains 25mg CBD and 25mg THC.
  Arms: Arm 3. Balanced arm (MPL-009)

SUMMARY:
CANnabinoids in Pediatric ONCology is a randomized, double blind, adaptive clinical trial looking at the tolerability of cannabinoids in children with cancer across 3 Canadian children's hospitals.

DETAILED DESCRIPTION:
This is a multi-centered, pragmatic, double-blind, adaptive, dose-escalation study to establish the tolerability of Cannabis Herbal Extracts (CHE) containing different ratios of delta-9 tetrahydrocannabinol (THC) and cannabidiol (CBD). Study arms will contain the following ratios THC:CBD 1:25 (arm 1), 1:5 (arm 2) and 1:1 (arm 3). CAN-PONC will enroll 20 participants recruited into each arm, for a total of 60 study participants.

To inform the dose for the arm containing the most THC, this study will take place in two stages. In Stage One: The first 20 participants will be randomized 1:1 into arm 1 and arm 2. Once 20 participants have been recruited, trial recruitment will halt until the last participant reaches the maintenance phase, the maximum THC dose at which less than 30% of participants reported dose limiting toxicities (Max-D30) has been established, the remaining 40 recruited participants will be randomized 1:1:2 into arm 1, arm 2 and arm 3 in Stage Two of this study.

All arms consist of three phases: baseline phase (no interventional product for two weeks), treatment phase (dose escalations for eight weeks), and a maintenance phase (maximum tolerated dose for four weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Ages 4-17 years old at the time of enrollment
2. Diagnosed with relapsed or refractory solid or hematologic malignancy including brain tumours
3. Currently receiving active cancer treatment or supportive and palliative care
4. Estimated survival of at least 4 months at the time of enrollment

Exclusion Criteria:

1. History of cardiovascular disease, severe hepatic or renal impairment defined by alanine transaminase (ALT)/ aspartate aminotransferase (AST) more than 5x upper limit of normal (ULN), creatinine more than 5x ULN or glomerular filtration rate (GFR less than) <60 mL/min/1.73 m273m2, unstable/unmanaged arrhythmias, uncontrolled hypertension with blood pressure above 99th centile for age or history of myocardial infarction
2. Nabilone or other cannabis-based products use (including for recreational purposes) within the past 2 weeks or planned nabilone use for the duration of their enrollment in the trial. Current use/continued use of recreational cannabis, or not willing to abstain from recreational cannabis use during the trial
3. Anyone who is pregnant or breast/chest-feeding throughout the duration of the study or has the intention to become pregnant within 3 months of study completion
4. Participation in other clinical trials that prohibit the concurrent use of cannabis
5. Children with a personal or family history of schizophrenia or psychotic disorders, substance use disorder or allergy to cannabinoids or cannabis
6. Unwilling or unable to use effective form of contraception and refrain from driving motorized vehicles (cars, motorcycles, boats, etc.) throughout the study period
7. Anyone who is currently receiving cell therapies or immune checkpoint inhibitors

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (Tolerability) | 14 weeks
  Reported through study completion

SECONDARY OUTCOMES:
Pain intensity | daily for 14 weeks
  Pain will be measured using Faces Pain Scale-Revised reported by the participants daily throughout the study. Pain will be reported for each study visit as a percentage change from the weekly average documented at baseline.
Symptom burden | 3 times per week for 14 weeks
  Symptom burden is measured using the score of Symptom Screening in Pediatrics Tool (SSPedi) assessed three times a week throughout the study and will be reported as a weekly average and percentage change from baseline.
Quality of life (child) | once per week for 14 weeks
  Pediatric quality of life inventory (PedsQLTM) will be assessed weekly throughout the study
Sleep (hours per night) | daily for 14 weeks
  Sleep, will be reported as the number of hours per night, measured using Actigraphy and/or parent report, will be reported as an average over a one-week time period.

CONTACTS AND LOCATIONS:
Overall Officials: Rod Rassekh, MD, Principal Investigator — University of British Columbia; Bruce Crooks, MD, Principal Investigator — Dalhousie University; Adam Rappoport, MD, Principal Investigator — The Hospital for Sick Children

IPD SHARING:
Plan to Share IPD: Undecided
No. Summary level data may be available from the CAN-PONC steering committee following research ethics board approval.